CLINICAL TRIAL: NCT05536245
Title: Analysis of the Prevalence of Violence Suffered or Committed by Patients Suffering From Addiction in a Care Facility
Acronym: APREVIO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2021 /PP-01
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Addictology
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — To prevalence of psychological, physical and sexual violence suffered or committed in a population of patients suffering from one or more addictions

SUMMARY:
Addictions, whether to a substance or a behavior, are often associated with violence, but their role is not well known. Despite the publication of numerous studies demonstrating the influence of addictions in acts of violence, the exploration of violence in the context of addiction remains very limited. In order to fill this gap, teams members of the Addictopôle Occitanie in collaboration with a regional team are preparing the launch of a concrete longitudinal study to analyze the incidence of violence in populations suffering from addiction, but also to evaluate the need in terms of management of this violence.

Hypotheses: To analyze the prevalence of violence in populations suffering from addiction and the need for treatment of such violence using a robust protocol based on an anonymous questionnaire to assess the violence experienced or committed by a patient, taking into account his/her environment. This study would allow us to better understand the effects of addictions on the severity and frequency of violence, but also to implement concrete and adapted solutions in order to limit it. This study could lead to the creation of a regional Observatory of Violence related to Addictions.

Translated with www.DeepL.com/Translator (free version)

DETAILED DESCRIPTION:
Study visits will be conducted in the following chronological order:

i. Inclusion/End Visit (IEV): D0.Eligible patients will have been identified by the investigator, and will be recruited in the Addictology Department during their usual visit.

The inclusion visit is carried out by an investigating physician who will confirm the patient's eligibility and verify his or her ability to answer the questionnaire. It will take place in the care center. It is part of the usual care.

During this visit, the investigator will:

* Perform the usual management of the patient.
* Validate the inclusion and non-inclusion criteria.
* Issue the letter of information and non-opposition

ii. Self-questionnaire entry visit (Vfollow-up/end): from D0 to 18 months (part of the usual care). After inclusion, the subject has enough time (15-30 min) to fill in the questionnaire independently. If the subject asks for it, the doctor can give him an explanation or clarify the meaning of a question and let him answer it alone. After completing the questionnaire, the subject will have no further obligations in relation to the study.The patient will complete an electronic self-questionnaire independently.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient under care in an Addictology structure.
* Male or female patient over 18 years old.
* Outpatient able to express his/her non-opposition.

Exclusion Criteria:

Patient consulting for the first time. Patient under court protection, guardianship or curatorship. Severe psychiatric disorders that have not been stabilized: (schizophrenia, bipolar disorders, etc.).

Severe neurological disorders that are incompatible with reliable data collection.

Minor patients. Pregnant women, parturients. People in emergency situations, people unable to express their consent.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients (stabilized out of crisis or under the influence of substances), men or women over 18 years of age who are able to understand the information letter and the questionnaire and to express their non-opposition. These patients must be under the care of an Addictology structure for addictive behavior, misuse of narcotics or for the consolidation of a sobriety
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Rate of violence among patients suffering from one or more addictions and treated in an Addictology Center. | Between Day1 and 18 Months
  Frequency of each type of violent act.

SECONDARY OUTCOMES:
Relation between addiction habits and violence | Between Day 1 and 18 Months
  Number of positive responses
Percentage of positive respons in terms of frequency of violence and need for specific help.and the acceptability of specific help by patients | Between Day 1 and 18 Months
  Number of positive responses

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Gaëlle SULTAN-TIHLL, Béziers
  - Hélène DONNADIEU, Montpellier
  - Pascal PERNEY, Nîmes
  - Nicolas FRANCHITTO, Toulouse